CLINICAL TRIAL: NCT04091542
Title: Hyperventilation and Oxygenation to Prolong Breath Hold in Breast Cancer Irradiation Treatment (HOBBIT): Development of Support Technique to Prolong Breath Hold Time During Radiotherapy
Brief Title: Hyperventilation and Oxygenation to Prolong Breath Hold in Breast Cancer Irradiation Treatment
Acronym: HOBBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC2019/0127
Record Dates: First submitted 2019-03-22; First posted 2019-09-16 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breath hold; hyperventilation; oxygenation
MeSH Terms: conditions — Breast Neoplasms; Hyperventilation | interventions — Ventilators, Mechanical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- FiO2 group 1 (Experimental): FiO2 changes over the four days in 60 with ventilator, 80 with ventilator, 60 with optiflow and 80 with optiflow.
  Interventions: Device: Optiflow/Ventilator
- FiO2 group 2 (Experimental): FiO2 changes over the four days in 80 with ventilator, 60 with ventilator, 80 with optiflow and 60 with optiflow.
  Interventions: Device: Optiflow/Ventilator
- Duration 1 (Experimental): In duration goup changes the preparation over the four days in 2 min. with ventilator, 6 min. with ventilator, 2 min. with optiflow and 8 min. with optiflow.
  Interventions: Device: Optiflow/Ventilator
- Duration 2 (Experimental): In duration goup changes the preparation over the four days in 6 min. with ventilator, 2 min. with ventilator, 6 min. with optiflow and 2 min. with optiflow.
  Interventions: Device: Optiflow/Ventilator
- respiratory rate 1 (Experimental): In the RR group changes the respiratory rate in the four days: 16 times with ventilator, 20 times with ventilator, 16 times with optiflow and 20 times with optiflow.
  Interventions: Device: Optiflow/Ventilator
- respiratory rate 2 (Experimental): In the RR group changes the respiratory rate in the four days: 20 times with ventilator, 16 times with ventilator, 20 times with optiflow and 16 times with optiflow.
  Interventions: Device: Optiflow/Ventilator
- Position 1 (Experimental): The position changes over the four days in supine with ventilator, prone with ventilator, supine with optiflow and prone with optiflow.
  Interventions: Device: Optiflow/Ventilator
- Position 2 (Experimental): The position changes over the four days in prone with ventilator, supine with ventilator, prone with optiflow and supine with optiflow.
  Interventions: Device: Optiflow/Ventilator

INTERVENTIONS:
Device: Optiflow/Ventilator — Participants will have 2 days with optiflow, 2 days with ventilator.

SUMMARY:
With the HOBBIT trial, the investigators want to develop a technology that allows volunteers to hold their breath for a long time. This technique will then be taught to patients with breast cancer to be able to hold their breath long-term during the irradiation. After all, research has shown that the heart is in a better position when the patient enters her breath after a deep inhalation, as a result of which there is less unwanted radiation of the heart. To develop this technique the investigators use healthy volunteers, who are asked several times to hold their breath as long as comfortable. Before the respiratory arrest the investigators allow these volunteers to hyperventilate, administer oxygen and cause hyperinflation of the lungs.

The volunteers come back four times, on four consecutive days. The first day they receive a short training. Afterwards oxygen is administered for a few minutes while the volunteers are asked to hyperventilate. Afterwards, by using the learned technique, they must hold their breath for as long as possible, comfortably. They should hold their breath 3 times in total with a short break in between. The following days there is always a change in the preparation protocol, compared to the previous study. Different parameters in the protocol will be changed for different groups of volunteers, this is based on randomization. In this way the effect of different parameters in the preparation of the AHS can be investigated. The investigators will use this information to develop a new protocol for extending the duration of breathing to two minutes and thirty seconds for use during radiotherapy treatment. The method for finding the optimal technique is iterative optimization. This method follows a process of development, testing, feedback and redevelopment cycles. Iteratively, these cycles of development use the prior research to further elaborate the most promising discoveries and drop paths that do not produce the desired result. During the development The investigators listen to the input of different people: doctors, nurses, support staff, engineers and the participants, to guarantee the usability of the technique on the radiotherapy device. Once the researchers think they have found a solution that meets all the conditions, a group of untrained volunteers are asked to implement the technique. With this the investigators validate the technique for later use in breast cancer patients.

DETAILED DESCRIPTION:
Radiotherapy (RT) has an established role in breast cancer, complementing surgery and systemic therapies to prevent recurrences and improve survival. Long-Term follow-up shows that the beneficial effect on survival is weakened by radiation-induced cardiac and lung cancer mortality, especially in patients with left sided breast cancer or requiring irradiation of regional lymph nodes. Cardiac toxicity is of major concern because many patients receive cardiotoxic systemic treatments like anthracyclines and trastuzumab. Dose and volume of the heart exposed to radiation correlate with severity of cardiac toxicity. The heart dose-volume parameters are highest for patients receiving left-side radiotherapy especially if irradiation of the internal mammary lymph nodes is performed. Risk of (fatal) ischemic heart attack increases linearly with mean heart dose with no known dose threshold. In patients who receive left-side local treatment, heart dose is decreased by using prone positioning or deep-inspiration breath hold (DIBH), or a combination of both.

Previous research has shown that the heart shifts to an anatomical more favorable position in DIBH, away from the breast, chest wall and internal mammary lymph nodes, reducing heart dose. This advantage remains in prone positioning. The goal is to prolong the duration of a single DIBH, to create a long-DIBH (L-DIBH). Possible advantages are better positioning of the patient, execution of technically more difficult procedures and inclusion of regional lymph node (locoregional) irradiation. Most patients can't sustain a DIBH long enough to perform simulation with computed tomography (CT) and delineation during DIBH, so delineation of the laser lines during CT-simulation is performed on the shallow breathing (SB) scan. During positioning of the patient on the radiotherapy machine, a daily cone-beam CT (CBCT) is performed. The duration of this CBCT is 40 seconds, maintaining DIBH during this period is also hard for most patients. So currently the positioning at the moment of treatment is based on the SB CT-scan, whilst the DIBH CT-scan is used for treatment. This could potentially induce suboptimal positioning. Breath hold during CBCT positioning and CT-simulation and delineation could minimize shifts in treatment position. The current DIBH schedules for whole breast cancer radiotherapy without inclusion of the lymph nodes, use between three and six DIBHs of 12 to 18 seconds. Longer DIBH could lead to less DIBHs and faster treatment execution, which is especially important when the lymph nodes are included in the target volumes. Locoregional irradiation, including the lymph nodes, requires between 10 and 14 DIBHs of 15-30 seconds which leads to a total treatment time of around 5 minutes. This represents a substantial physical and mental effort for all but the most able patients.

This research, the first phase of the Hyperventilation Oxygenation Breath hold in Breast cancer Irradiation Treatment (HOBBIT) trail, will focus on finding a technique to assist patients to maintain a long DIBH (L-DIBH) during radiotherapy. Other research has shown a potential increase in duration of breath hold and reduction in rest time between DIBHs using oxygen in combination with hyperventilation. There is a safe way to prolong DIBH to at least 5 minutes. However, the technique requires a long training period for the patient, and 15 minutes of mechanical ventilation before each treatment session, making the technique very time consuming and resource intensive. The investigators hope to simplify the technique by allowing patients to do multiple L-DIBHs during the 5 minutes of treatment time. The investigators found from preliminary tests that using shorter L-DIBHs has several advantages, firstly pre-oxygenation and induction of hypocapnia can be achieved in a shorter time, secondly the duration of training is reduced, and thirdly a the costs are reduced.

Increase in blood pressure is the main risk of L-DIBH. No adverse events of L-DIBH have been reported. In order to minimize the risks during testing, this research project was developed in collaboration with the anesthesiology department, to ensure safety of the participants during L-DIBH. For all subjects, vital parameters will be continuously monitored by medical staff. Safety boundaries are in place which subjects are not allowed to cross during L-DIBH.

The aim of this research is to develop a new and easy technique for L-DIBH in prone and supine position, feasible for daily use at our radiotherapy department. The purpose of the technique is to allow locoregional treatment using a reasonable amount of L-DIBHs, increase patient positioning and accuracy of radiation treatment, and further significantly reduce heart toxicity for left sided cancer patients. The HOBBIT trial includes multiple phases. The first phase is performed on healthy volunteers, different support techniques to prolong DIBH will be tested. In the second phase the most optimal techniques to perform a L-DIBH will be validated on breast cancer patients. Around 40 volunteers will be included in the first phase of the HOBBIT trail, the final amount of volunteers depends on the amount of testing needed to find a technique which fulfills all criteria for phase two. The second phase of the HOBBIT trail will include breast cancer patients treated at our radiotherapy center. The expectations from previous research is that the investigators will see a similar increase in DIBH time, compared to healthy volunteers. The final goal is the use of the technique during locoregional radiation therapy at the University Hospital of Ghent.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Volunteer
* Age ≥ 18 years
* Karnofsky index of at least 90
* Single DIBH of at least twenty seconds without assistance
* Informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* Pregnant women
* Volunteers above WHO Obesity class II (BMI>35kg/m²)
* Subjects on oxygen treatment during day or night
* COPD or Asthma patients
* Volunteers with pulmonary hypertension
* New York Heart Association functional classification (NYHA) of 2 or less
* Personal history of cerebrovascular disease, aortic disease, coronary artery disease or myocardial disease
* Treatment with antihypertensive medication
* Missing more than three teeth without use of a prosthesis
* Gastric tube present
* Smoking
* Previous breath-holding experience (e.g. diver, etc.)
* Anxiety symptoms grade 1 or higher according to CTCAE v.5
* Mental condition rendering the volunteer unable to understand the nature, scope and possible consequences of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
conditions for a technique for L-DIBHs of more than two minutes thirty seconds | 2 years
  duration of preparation/hyperventilation and oxygenation

SECONDARY OUTCOMES:
Oxygen saturation | 1 year
  fraction of [oxygen]-saturated hemoglobin relative to total hemoglobin in the blood
heart rate | 1 year
  speed of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm)
diastolic and systolic blood pressure | 1 year
  the pressure of circulating blood on the walls of blood vessels
EtCO2 | 1 year
  patient's end-tidal CO2
average L-DIBH time | 1 year
  measured in minutes and seconds
average time needed for SpO2 to recover to normal | 1 year
  measured in minutes and seconds
average total time needed to perform three L-DIBHs consequently | 1 year
  measured in minutes and seconds
Measurement of linear anteroposterior displacement | 1 year
  measured in millimetres
dizziness | 1 year
  an impairment in spatial perception and stability.
fear | 1 year
  a feeling induced by perceived danger or threat that occurs in certain types of organisms, which causes a change in metabolic and organ functions and ultimately a change in behavior, such as fleeing, hiding, or freezing from perceived traumatic events
headache | 1 year
  the symptom of pain anywhere in the region of the head or neck
syncope | 1 year
  syncope
coughing | 1 year
  a sudden, and often repetitively occurring, protective reflex which helps to clear the large breathing passages from fluids, irritants, foreign particles and microbes
dyspnea | 1 year
  the feeling that one cannot breathe well enough
nausea | 1 year
  an unpleasant, diffuse sensation of unease and discomfort, often perceived as an urge to vomit
vomiting | 1 year
  the involuntary, forceful expulsion of the contents of one's stomach through the mouth and sometimes the nose
itching | 1 year
  a sensation that causes the desire or reflex to scratch
pain | 1 year
  a distressing feeling often caused by intense or damaging stimuli
palpitations | 1 year
  the perceived abnormality of the heartbeat characterized by awareness of cardiac muscle contractions in the chest, which is further characterized by the hard, fast and/or irregular beatings of the heart
blurred vision | 1 year
  an ocular symptom
muscle cramps | 1 year
  a sudden, involuntary muscle contraction or over-shortening; while generally temporary and non-damaging, they can cause significant pain, and a paralysis-like immobility of the affected muscle

CONTACTS AND LOCATIONS:
Overall Officials: Liv Veldeman, dr, Principal Investigator — University Ghent
Locations (1):
- University Hospital - Radiotherapy Department, Ghent, Belgium